CLINICAL TRIAL: NCT05964790
Title: A Phase Ⅰb/Ⅱ, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Investigate the Safety, Tolerability, Pharmacokinetics and Efficacy of HS-10380 in Chinese Adults With Schizophrenia.
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy Study of HS-10380 in Patients With Schizophrenia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-10380-201
Record Dates: First submitted 2023-07-10; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Psychotropic drug; Antipsychotic agents
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10380 (Experimental): Participants received HS-10380 tablet orally once daily for 28 days.
  Interventions: Drug: HS-10380
- Placebo (Placebo Comparator): Participants received placebo tablet matching HS-10380 1.5mg tablet orally once daily for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HS-10380 — Participants in arm HS-10380 will receiving multiple ascending doses of HS-10380 (1.5 mg initial dose) orally once daily for 28 days
  Arms: HS-10380
Drug: Placebo — Participants in arm Placebo will receiving multiple ascending doses of Placebo matching HS-10380 (1.5 mg initial dose) orally once daily for 28 days
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, pharmacokinetics and efficacy of HS-10380 relative to placebo for the treatment of participants with schizophrenia.

DETAILED DESCRIPTION:
The trial consists of two parts: dose escalation cohorts and expansion cohorts. The primary aim of the dose escalation cohorts is to evaluate the safety and tolerability of HS-10380 in participants with schizophrenia, and the primary aim of expansion cohorts is to evaluate efficacy of HS-10380 in participants with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation cohorts:

  1. Patients are 18 to 55 years of age, inclusive.
  2. Body mass index (BMI) between 18.5 and 30.0 kg/m2 ,inclusive. Weight ≥ 50 kg for male subjects and ≥ 45 kg for female subjects.
  3. Patient meets DSM-5 criteria for schizophrenia.
  4. Currently not taking antipsychotics. Or on a stable dose of single second-generation antipsychotics (SGA) for at least 2 weeks, limited to either risperidone, olanzapine, quetiapine, aripiprazole, or paliperidone.
  5. PANSS total score ≤ 90. Rating ≤ 4 on hostility and uncooperativeness,
  6. Negative urine pregnancy test (women of childbearing potential only).
  7. Male and female patients must agree to use a highly effective method of birth control during the course of the entire study and for 3 months after the last dose of investigational product.
  8. Written informed consent has been obtained.

Expansion cohorts:

1. Patients are 18 to 65 years of age, inclusive.
2. Patient meets DSM-5 criteria for schizophrenia.
3. No current use of antipsychotics. Or withdrawing from antipsychotics other than clozapine for more than 5 half-lives prior to randomization.
4. PANSS total score ≥70 and ≤120. Rating of at least 4 (moderate) on at least 2 of the following 4 PANSS positive symptoms; P1: delusions; P2: conceptual disorganization; P3: hallucinatory behavior; P6: suspiciousness/persecution.
5. Negative urine pregnancy test (women of childbearing potential only).
6. Male and female patients must agree to use a highly effective method of birth control during the course of the entire study and for 3 months after the last dose of investigational product.
7. Written informed consent has been obtained.

Exclusion Criteria:

* Dose escalation cohorts:

  1. Patients meet DSM-5 criteria for a mental illness other than schizophrenia, and might interfere with the conduct of the study as determined by the investigator.
  2. Current risk of self-harm or violence, including: having any suicidal ideation or suicidal behavior within the last 6 months, as assessed using Columbia-Suicidal Severity Rating Scale (C-SSRS).
  3. Patients who have a clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorder, etc. Medical conditions that are minor or well-controlled may be considered acceptable if the condition does not interfere with the conduct of the study.
  4. Patients who received electroconvulsive therapy (ECT) within 3 months prior to screening.
  5. Received a long-acting antipsychotic within 6 months prior to screening or within the duration of 5 half-lives of the drug.
  6. History of seizure disorder (with the exception of febrile seizure).
  7. History of malignant syndrome.
  8. Any condition that would be expected to affect drug absorption, distribution, metabolism and excretion, including gastrointestinal surgery, urinary tract obstruction or difficulty in urination, etc.
  9. History of severe allergies.
  10. Female patients who are pregnant, puerperal or breastfeeding.
  11. History of drug addiction within 1 year prior to screening.
  12. Patients who has a history of alcohol abuse (defined as more than 14 standard units of alcohol consumption per week, 1 standard unit = 360 mL of beer, 45 mL of distilled spirits or 150 mL of wine) within 6 months prior to screening, or are unable to abstain from alcohol use during the study period.
  13. Patients who smoke ≥10 cigarettes per day within 3 months prior to screening, or are unable to quit smoking during the study period.
  14. Abnormal physical examination results that may interfere with the study.
  15. Abnormal vital signs that may interfere with the study, including: resting heart rate <60 or >100 beats per minute, systolic blood pressure <90mmHg or ≥140mmHg, diastolic blood pressure <60mmHg or ≥90mmHg.
  16. Abnormal electrocardiogram (ECG) results may interfere with the study, including: QTcF>450ms for male subjects and >470ms for female subjects based on Fridericia correction.
  17. Abnormal clinical laboratory test results may interfere with the study, including: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) results >1.5 × the upper limit of normal (ULN); serum prolactin levels >5 × ULN or significant clinical symptoms like amenorrhea, gynecomastia, and lactation.
  18. Patients whose results for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), or syphilis serological reaction (TRUST) is not negative.
  19. Blood donation or blood loss ≥ 200ml within 1 month prior to screening.
  20. Patients requiring concomitant treatment with a moderate or strong cytochrome P450 (CYP) 3A4 inhibitors or CYP3A4 inducers, or a moderate or strong cytochrome CYP2D6 inhibitors or CYP3A4 inducers.
  21. Prior participation in any Interventional clinical trials within 3 months.
  22. Unsuitable for any other reason, as judged by the investigator.

Expansion cohorts:

1. Patients meet DSM-5 criteria for a mental illness other than schizophrenia, and might interfere with the conduct of the study as determined by the investigator.
2. Current risk of self-harm or violence, including: having any suicidal ideation or suicidal behavior within the last 6 months, as assessed using Columbia-Suicidal Severity Rating Scale (C-SSRS).
3. Patients who have a clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorder, etc. Medical conditions that are minor or well-controlled may be considered acceptable if the condition does not interfere with the conduct of the study.
4. Patients who received electroconvulsive therapy (ECT) within 3 months prior to screening.
5. Received a long-acting antipsychotic within 6 months prior to screening or within the duration of 5 half-lives of the drug.
6. History of seizure disorder (with the exception of febrile seizure).
7. History of malignant syndrome.
8. Any condition that would be expected to affect drug absorption, distribution, metabolism and excretion, including gastrointestinal surgery, urinary tract obstruction or difficulty in urination, etc.
9. History of severe allergies.
10. Female patients who are pregnant, puerperal or breastfeeding.
11. History of drug addiction within 1 year prior to screening.
12. Patients who has a history of alcohol abuse (defined as more than 14 standard units of alcohol consumption per week, 1 standard unit = 360 mL of beer, 45 mL of distilled spirits or 150 mL of wine) within 6 months prior to screening, or are unable to abstain from alcohol use during the study period.
13. Abnormal physical examination results that may interfere with the study.
14. Abnormal vital signs that may interfere with the study, including: resting heart rate <60 or >100 beats per minute, systolic blood pressure <90mmHg or ≥140mmHg, diastolic blood pressure <60mmHg or ≥90mmHg.
15. Abnormal electrocardiogram (ECG) results may interfere with the study, including: QTcF>450ms for male subjects and >470ms for female subjects based on Fridericia correction.
16. Abnormal clinical laboratory test results may interfere with the study, including: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) results > 2 × the upper limit of normal (ULN).
17. Patients whose results for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), or syphilis serological reaction (TRUST) is not negative.
18. Patients requiring concomitant treatment with a moderate or strong cytochrome P450 (CYP) 3A4 inhibitors or CYP3A4 inducers, or a moderate or strong cytochrome CYP2D6 inhibitors or CYP3A4 inducers.
19. Blood donation or blood loss ≥ 200ml within 1 month prior to screening.
20. Prior participation in any Interventional clinical trials within 3 months.
21. Unsuitable for any other reason, as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose escalation cohorts: Incidence and severity of adverse events(AE) ，serious AEs and AE leading to withdrawal from treatment. | Baseline to Day 43
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A serious AE (SAE) is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or is a congenital anomaly/birth defect.
Dose escalation cohorts: Changes from baseline in complete blood count (CBC). | Baseline to Day 36
  Hematology parameters to be reported: white blood cells, red blood cells and platelets.
Dose escalation cohorts: Changes from baseline in urinalysis. | Baseline to Day 36
  Parameters to be reported: protein, glucose, ketones, red blood cells, and white blood cells.
Dose escalation cohorts: Changes from baseline in blood biochemistry test. | Baseline to Day 36
  Parameters to be reported: glucose, urea, serum creatinine, alanine aminotransferase, aspartate transaminase, albumin, total protein, bilirubin, and blood lipid index.
Dose escalation cohorts: Changes from baseline in coagulation function test. | Baseline to Day 36
  prothrombin time, activated partial thromboplastin time and international normalized ratio.
Dose escalation cohorts: Changes from baseline in thyroid function test. | Baseline to Day 36
  thyroxine, triiodothyronine, free triiodothyronine, free thyroxin and thyroid stimulating hormone.
Dose escalation cohorts: Changes from baseline in serum prolactin. | Baseline to Day 36
  Laboratory test.
Dose escalation cohorts: Changes from baseline in blood pressure (BP). | Baseline to Day 36
  Vital sign.
Dose escalation cohorts: Changes from baseline in pulse rate. | Baseline to Day 36
  Vital sign.
Dose escalation cohorts: Changes from baseline in body temperature. | Baseline to Day 36
  Vital sign.
Dose escalation cohorts: Change from baseline in body weight | Baseline to Day 29
  Body weight was measured in kilograms (Kg).
Dose escalation cohorts: Change from baseline in Electrocardiogram (ECG) | Baseline to Day 36
  ECG parameters including heart rate, PR interval, RR interval and QTcF, etc.
Dose escalation cohorts: Change from baseline in Simpson-Angus Scale (SAS) | Baseline to Day 36
  SAS is a 10-item testing instrument used to evaluate drug-related extrapyramidal syndromes. The following items are included in the SAS: gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head dropping, glabella reflex, tremor, and salivation. Total score ranges from 0 to 40 with a higher score indicating increased severity.
Change from baseline in Abnormal Involuntary Movement Scale (AIMS) | Baseline to Day 36
  AIMS is a rating scale measuring involuntary movements known as tardive dyskinesia, that sometimes develop as a side effect of long-term treatment with antipsychotic medications. The AIMS score was calculated as the sum of questions 1 through 7 of the AIMS instrument, which includes assessments of involuntary movements in the face, lips, jaw, tongue, upper and lower extremities, and neck/shoulders/hips. Each item is rated on a five-point scale of severity from 0-4 with 0 (none), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe). Total scores range from 0 to 28.
Dose escalation cohorts: Change from baseline in Barnes Akathisia Rating Scale | Baseline to Day 36
  BARS is a rating scale that is administered by physicians to assess the severity of drug-induced akathisia, which is a movement disorder characterized by a feeling of inner restlessness and a compelling need to be in constant motion, as well as by actions such as rocking while standing or sitting, lifting the feet as if marching on the spot, and crossing and uncrossing the legs while sitting. The following subcategories are scored: objective akathisia, subjective awareness of restlessness and subjective distress related to restlessness and are rated on a 4-point scale from 0-3. In addition, the global clinical assessment of akathisia uses a 6-point scale ranging from 0-5. Total score ranges from 0 to 14 with a higher score indicating increased severity.
Dose escalation cohorts: Change from Baseline in Columbia - Suicide Severity Rating Scale (C-SSRS) | Baseline to Day 36
  C-SSRS is a scale capturing occurrence, severity, and frequency of suicide-related thoughts and behaviors, and has a binary response (yes/no). Suicidal Ideation: a "yes" answer to any one of 5 suicidal ideation questions: Wish to be Dead, Non-specific Active Suicidal Thoughts, Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act, Active Suicidal Ideation with Some Intent to Act, without Specific Plan, Active Suicidal Ideation with Specific Plan and Intent. Suicidal Behavior: a "yes" answer to any of 5 suicidal behavior questions: Preparatory Acts or Behavior, Aborted Attempt, Interrupted Attempt, Actual Attempt (non-fatal), Completed Suicide.
Expansion cohorts: Change from Baseline in Positive and Negative Syndrome Scale (PANSS) | Baseline to Day 28
  PANSS is a 30-item rating scale specifically developed to asses both the positive and negative symptom syndromes of patients with schizophrenia. PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210. Higher PANSS total score means more severe outcome.
Expansion cohorts: Positive and Negative Syndrome Scale (PANSS) Response at Week 4, Defined as a 20% or Greater Improvement from Baseline in PANSS Total Score | Baseline to Day 28
  PANSS is a 30-item rating scale specifically developed to asses both the positive and negative symptom syndromes of patients with schizophrenia. PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210. Higher PANSS total score means more severe outcome.
Expansion cohorts: Change from Baseline in Clinical Global Impression-Severity (CGI-S) | Baseline to Day 28
  CGI-S is a clinician-rated scale that measures the overall severity of a participant's illness in comparison with the severity of illness in other participants the physician has observed.
  The CGI-S a single-item clinician-rated assessment of the subject's current illness state on a 7-point scale (score range: 1-7), where a higher score is associated with greater illness severity.

SECONDARY OUTCOMES:
Dose escalation cohorts: Maximum plasma concentration (Cmax) of first HS-10380 administration | Baseline to Day 36
  Pharmacokinetics describes the action of a drug in the body over a period of time. Blood samples are collected to measure plasma concentrations of the study drug at different times after dosing.
Dose escalation cohorts: Time of the Maximum Concentration (Tmax) of first HS-10380 administration | Baseline to Day 36
  Pharmacokinetics describes the action of a drug in the body over a period of time. Blood samples are collected to measure plasma concentrations of the study drug at different times after dosing.
Dose escalation cohorts: Area under the concentration time curve of intervals (AUC0-τ) of first HS-10380 administration | Baseline to Day 36
  Pharmacokinetics describes the action of a drug in the body over a period of time. Blood samples are collected to measure plasma concentrations of the study drug at different times after dosing.
Dose escalation cohorts: Area under the concentration time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC0-t) of first HS-10380 administration | Baseline to Day 36
  Pharmacokinetics describes the action of a drug in the body over a period of time. Blood samples are collected to measure plasma concentrations of the study drug at different times after dosing.
Dose escalation cohorts: Maximum concentration at steady state (Css, max) of multiple-dose HS-10380 administration | Baseline to Day 36
  Pharmacokinetics describes the action of a drug in the body over a period of time. Blood samples are collected to measure plasma concentrations of the study drug at different times after dosing.
Dose escalation cohorts: Time of the maximum concentration at steady state (Tss, max) of multiple-dose HS-10380 administration | Baseline to Day 36
  Pharmacokinetics describes the action of a drug in the body over a period of time. Blood samples are collected to measure plasma concentrations of the study drug at different times after dosing.
Dose escalation cohorts: Minimum concentration at steady state (Css, min) of multiple-dose HS-10380 administration | Baseline to Day 36
  Pharmacokinetics describes the action of a drug in the body over a period of time. Blood samples are collected to measure plasma concentrations of the study drug at different times after dosing.
Dose escalation cohorts: Area under the concentration-time curve at steady state (AUCss) of multiple-dose HS-10380 administration | Baseline to Day 36
  Pharmacokinetics describes the action of a drug in the body over a period of time. Blood samples are collected to measure plasma concentrations of the study drug at different times after dosing.
Dose escalation cohorts: Apparent clearance at steady state (CLss/F) of multiple-dose HS-10380 administration | Baseline to Day 36
  Pharmacokinetics describes the action of a drug in the body over a period of time. Blood samples are collected to measure plasma concentrations of the study drug at different times after dosing.
Dose escalation cohorts: Apparent volume of distribution at steady state (Vss/F) of multiple-dose HS-10380 administration | Baseline to Day 36
  Pharmacokinetics describes the action of a drug in the body over a period of time. Blood samples are collected to measure plasma concentrations of the study drug at different times after dosing.
Dose escalation cohorts: Change from Baseline in Positive and Negative Syndrome Scale (PANSS) | Baseline to Day 28
  PANSS is a 30-item rating scale specifically developed to asses both the positive and negative symptom syndromes of patients with schizophrenia. PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210. Higher PANSS total score means more severe outcome.
Dose escalation cohort: Positive and Negative Syndrome Scale (PANSS) Response at Week 4, Defined as a 20% or Greater Improvement from Baseline in PANSS Total Score | Baseline to Day 28
  PANSS is a 30-item rating scale specifically developed to asses both the positive and negative symptom syndromes of patients with schizophrenia. PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210. Higher PANSS total score means more severe outcome.
Dose escalation cohorts: Change from Baseline in Clinical Global Impression-Severity (CGI-S) | Baseline to Day 28
  CGI-S is a clinician-rated scale that measures the overall severity of a participant's illness in comparison with the severity of illness in other participants the physician has observed.
  The CGI-S a single-item clinician-rated assessment of the subject's current illness state on a 7-point scale (score range: 1-7), where a higher score is associated with greater illness severity.
Expansion cohorts: Incidence and severity of adverse events(AE) ，serious AEs and AE leading to withdrawal from treatment. | Baseline to Day 43
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A serious AE (SAE) is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or is a congenital anomaly/birth defect.
Expansion cohorts: Changes from baseline in complete blood count (CBC). | Baseline to Day 36
  Hematology parameters to be reported: white blood cells, red blood cells and platelets.
Expansion cohorts: Changes from baseline in urinalysis. | Baseline to Day 36
  Parameters to be reported: protein, glucose, ketones, red blood cells, and white blood cells.
Expansion cohorts: Changes from baseline in blood biochemistry test. | Baseline to Day 36
  Parameters to be reported: glucose, urea, serum creatinine, alanine aminotransferase, aspartate transaminase, albumin, total protein, bilirubin, and blood lipid index.
Expansion cohorts: Changes from baseline in coagulation function test | Baseline to Day 36
  prothrombin time, activated partial thromboplastin time and international normalized ratio.
Expansion cohorts: Changes from baseline in hyroid function test | Baseline to Day 36
  thyroxine, triiodothyronine, free triiodothyronine, free thyroxin and thyroid stimulating hormone.
Expansion cohorts: Changes from baseline in serum prolactin | Baseline to Day 36
  Laboratory test.
Expansion cohorts: Changes from baseline in blood pressure (BP) | Baseline to Day 36
  Vital sign.
Expansion cohorts: Changes from baseline in pulse rate | Baseline to Day 36
  Vital sign.
Expansion cohorts: Changes from baseline in body temperature | Baseline to Day 36
  Vital sign.
Expansion cohorts: Change from baseline in body weight | Baseline to Day 29
  Body weight was measured in kilograms (Kg).
Expansion cohorts: Change from baseline in Electrocardiogram (ECG) | Baseline to Day 36
  ECG parameters including heart rate, PR interval, RR interval and QTcF, etc.
Expansion cohorts: Change from baseline in Simpson-Angus Scale (SAS) | Baseline to Day 36
  SAS is a 10-item testing instrument used to evaluate drug-related extrapyramidal syndromes. The following items are included in the SAS: gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head dropping, glabella reflex, tremor, and salivation. Total score ranges from 0 to 40 with a higher score indicating increased severity.
Expansion cohorts: Change from baseline in Abnormal Involuntary Movement Scale (AIMS) | Baseline to Day 36
  AIMS is a rating scale measuring involuntary movements known as tardive dyskinesia, that sometimes develop as a side effect of long-term treatment with antipsychotic medications. The AIMS score was calculated as the sum of questions 1 through 7 of the AIMS instrument, which includes assessments of involuntary movements in the face, lips, jaw, tongue, upper and lower extremities, and neck/shoulders/hips. Each item is rated on a five-point scale of severity from 0-4 with 0 (none), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe). Total scores range from 0 to 28.
Expansion cohorts: Change from baseline in Barnes Akathisia Rating Scale | Baseline to Day 36
  BARS is a rating scale that is administered by physicians to assess the severity of drug-induced akathisia, which is a movement disorder characterized by a feeling of inner restlessness and a compelling need to be in constant motion, as well as by actions such as rocking while standing or sitting, lifting the feet as if marching on the spot, and crossing and uncrossing the legs while sitting. The following subcategories are scored: objective akathisia, subjective awareness of restlessness and subjective distress related to restlessness and are rated on a 4-point scale from 0-3. In addition, the global clinical assessment of akathisia uses a 6-point scale ranging from 0-5. Total score ranges from 0 to 14 with a higher score indicating increased severity.
Expansion cohorts: Change from Baseline in Columbia - Suicide Severity Rating Scale (C-SSRS) | Baseline to Day 36
  C-SSRS is a scale capturing occurrence, severity, and frequency of suicide-related thoughts and behaviors, and has a binary response (yes/no). Suicidal Ideation: a "yes" answer to any one of 5 suicidal ideation questions: Wish to be Dead, Non-specific Active Suicidal Thoughts, Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act, Active Suicidal Ideation with Some Intent to Act, without Specific Plan, Active Suicidal Ideation with Specific Plan and Intent. Suicidal Behavior: a "yes" answer to any of 5 suicidal behavior questions: Preparatory Acts or Behavior, Aborted Attempt, Interrupted Attempt, Actual Attempt (non-fatal), Completed Suicide.

IPD SHARING:
Plan to Share IPD: No